CLINICAL TRIAL: NCT02612701
Title: E-Cigarette Aerosol, Conventional Cigarette Smoke, and Myocardial Perfusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the pandemic we decided to terminate this project.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Florian Rader, M.D, M.Sc., Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00041957
Record Dates: First submitted 2015-11-17; First posted 2015-11-24 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease; Myocardial Perfusion
Keywords: Myocardial perfusion; Electronic cigarettes; Cigarettes; Cigarette smoking
MeSH Terms: conditions — Coronary Artery Disease; Vaping; Cigarette Smoking | interventions — Tobacco Products; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cigarettes (Experimental): Healthy chronic dual cigarette and e-cigarette smokers will undergo myocardial contrast echocardiography before and after smoking two standard cigarettes
  Interventions: Other: Cigarettes
- E-cigarettes (nicotine free e-liquid) (Experimental): Healthy chronic dual cigarette and e-cigarette smokers will undergo myocardial contrast echocardiography before and after smoking nicotine free e-cigarette liquid.
  Interventions: Other: E-cigarettes (nicotine free e-liquid)
- E-cigarettes (low nicotine e-liquid) (Experimental): Healthy chronic dual cigarette and e-cigarette smokers will undergo myocardial contrast echocardiography before and after smoking low concentration(4-6 mg/mL) e-cigarette liquid.
  Interventions: Other: E-cigarettes (low nicotine e-liquid)
- E-cigarettes (high nicotine e-liquid) (Experimental): Healthy chronic dual cigarette and e-cigarette smokers will undergo myocardial contrast echocardiography before and after smoking high concentration (18-24 mg/mL) e-cigarette liquid.
  Interventions: Other: E-cigarettes (high nicotine e-liquid)

INTERVENTIONS:
Other: Cigarettes — Subjects will smoke a standard cigarette (yield: tar 12 mg, nicotine 1 mg)
  Arms: Cigarettes
Other: E-cigarettes (nicotine free e-liquid) — Subjects will smoke nicotine free e-liquid with an e-cigarette.
  Arms: E-cigarettes (nicotine free e-liquid)
Other: E-cigarettes (low nicotine e-liquid) — Subjects will smoke low nicotine (4-6 mg/mL) e-liquid with an e-cigarette.
  Arms: E-cigarettes (low nicotine e-liquid)
Other: E-cigarettes (high nicotine e-liquid) — Subjects will smoke low nicotine (18-24 mg/mL) e-liquid with an e-cigarette.
  Arms: E-cigarettes (high nicotine e-liquid)

SUMMARY:
E-cigarettes deliver nicotine by creating an aerosol of ultrafine particles. Many questions remain about the size and composition and especially about the potential toxicity of these particles. Thus, a key unanswered question-and the research question proposed-is whether e-cigarette aerosol triggers the same acute impairment in coronary microvessel function as does conventional cigarette smoke, which delivers a very well-defined exposure to fine particles and many fold greater exposure to toxic (combustion) products including volatile organic compounds (such as acrolein) that have been implicated in the pathogenesis of tobacco-related coronary disease.

Because the effects of nicotine on the human coronary microcirculation remain incompletely defined-with multiple potential vasodilator and vasoconstrictor actions each of which may vary by dose-we will determine the comparative effects of conventional cigarette smoke against e-cigarette aerosol with no nicotine, with low-dose nicotine, and with high-dose nicotine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49
* Regular cigarette smoker defined as at least 1 pack year and ≥ 5/day
* E-cigarette smoker defined as ≥ 1/week in the last 6 months.

Exclusion Criteria:

* Sub-optimal echocardiography images as determined by the sonographer and/or investigators.
* History of cardiopulmonary (including asthma or use of inhalers),
* History of diabetes or dyslipidemia
* History of psychiatric illness
* Blood Pressure > 140/90
* Body Mass Index ≤ 18.5 or ≥ 30 kg•m2
* Evidence of any of the above by physical examination, Electrocardiogram (ECG) or echocardiogram
* Resting Heart Rate > 100 beats/min
* Cardiac rhythm disorder, specifically: rhythm other than sinus, Supraventricular Tachycardia (SVT), atrial fibrillation, ventricular tachycardia
* Use of prescription medication except oral contraceptive pills
* History of illicit drug use (self-stated)
* Pregnant
* Any other condition(s) deemed by the physician investigators that put subjects at risk for participating in the study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-10-01 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Myocardial Perfusion (change in microvascular flux rate from baseline at 30 minutes) | Baseline and 30 minutes after smoking
  Myocardial contrast echocardiography will be used to measure regional myocardial perfusion - microvascular flux rate
Myocardial Perfusion (change in capillary blood volume from baseline at 30 minutes) | Baseline and 30 minutes after smoking
  Myocardial contrast echocardiography will be used to measure regional myocardial perfusion - capillary blood volume

CONTACTS AND LOCATIONS:
Overall Officials: Florian Rader, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States